CLINICAL TRIAL: NCT04101305
Title: Measurement of Circulating Tumor Cells in Prostate Cancer
Acronym: ICELLATEPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Karolinska Institutet (Other); iCellate Medical (Industry)
Responsible Party: Principal Investigator, Christer Ericsson, Senior scientist, Sormland County Council, Sweden
Other Study IDs: 2019-02592
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer, biomarker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Localised prostate cancer: Patients diagnosed with prostate cancer of moderate estimated risk suitable for and scheduled for prostatectomy with gland evacuation
  Interventions: Diagnostic Test: IsoPic
- Stage 3 prostate cancer: Patients with diagnosed stage 3 prostate cancer
  Interventions: Diagnostic Test: IsoPic
- Stage 4 prostate cancer: Patients with diagnosed stage 4 prostate cancer
  Interventions: Diagnostic Test: IsoPic
- Healthy controls: Age-matched healthy individuals free from diagnosed cancer, but with benign inflammatory prostatitis or other benign urological condition
  Interventions: Diagnostic Test: IsoPic

INTERVENTIONS:
Diagnostic Test: IsoPic — Biomimetic circulating epithelial cell enrichment followed by epithelial cell detection and single cell DNA sampling and sequencing

SUMMARY:
Can tumor cells and tumor DNA be sampled from blood samples from prostate cancer patients? Is it possible to understand the causal relationship between the occurrence of the tumor cells and the tumor DNA in the blood by reviewing the patient's medical records, including information about investigations, analytical reports or diagnoses? Can gene defects that may be useful in predicting the best treatment be detected by sequencing individual tumor cells or plasma from blood samples?

DETAILED DESCRIPTION:
Prostate cancer is the most common form of cancer in men and the second most deadly. Today's diagnostic methods and treatments are therefore obviously not adequate. In this study we will evaluate a new diagnostic sampling and analysis method for prostate cancer, not try new treatments. The test sampling involves the rare tumor cells and tumor DNA found in the blood, and sequencing their DNA to determine which, if any, defective genes they contain that may explain the disease. There is currently no universally accepted diagnostic test of either tumor cells or tumor DNA in blood. We have access to new technology that one of us (CE) developed at the Karolinska Institute, which by all accounts can give access to the rare tumor cells in the blood so that we can sequence their DNA. In this study we want to try to see if it is possible in practical healthcare to apply the new technology for prostate cancer patients and if there are signs that it works equally well in the healthcare environment as in the laboratory.

Impact: If the sampling of tumor cells and tumor DNA from blood samples works within the healthcare system processes, it will be possible to understand the causal relationships behind their occurrence, and their gene defects, we can design follow-up studies that would take us closer to clinical use of the new technology to predict which treatment would be most effective and which treatment would produce the least side effects.

Ethical considerations: The risks of blood sampling are limited and known and can be managed within the healthcare system. Data is handled safely. The potential future benefit of a new cancer cell- and DNA-test is great.

The study is a collaboration between Region Sörmland, Karolinska Institutet and iCellate Medical AB. The data collection is expected to be completed in 2020 and the analyses in 2021.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with prostate cancer of moderate risk planned for prostatectomy with lymph node removal, or
* patients diagnosed with prostate cancer stage 3, or
* patients with diagnosed prostate cancer stage 4, or
* patients with diagnosed benign inflammatory prostatitis or other benign urological condition constituting age-matched, cancer free, controls

Exclusion Criteria:

* Patients undergoing prostate cancer treatment (no prostate cancer treatment should be given to the patient before blood collection)
* Patients with previous malignancy

Ages: 18 Years to 125 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Study Population: Patients referred to the urology clinic for investigation of a suspected urologic condition
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Single cell DNA sampling | September 2019 to December 31st, 2020
  Can tumor cells and tumor DNA be sampled from blood samples from prostate cancer patients with various advanced disease?

SECONDARY OUTCOMES:
Comparison of novel sampling results to established biomarkers | September 2019 to December 31st, 2020
  Is it possible to understand the causal link between the presence and amounts of tumor cells and tumor DNA in the blood by reviewing the patient's medical records, including information on investigations, analysis reports and diagnosis?
Single cell DNA sequencing | September 2019 to December 31st, 2020
  Can acquired gene defects that may predict treatment be detected by sequencing individual tumor cells, or break-down products, from blood samples?

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Digkas, MD, PhD, Study Director — Region Sormland
Locations (1):
- Malarsjukhuset, Eskilstuna, Sormland, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Castro et al., Surgery Curr Res 2012, 2:3 http://dx.doi.org/10.4172/2161-1076.1000113
- [Background] Castro et al., J Integr Oncol 2018, 7:3 DOI: 10.4172/2329-6771.1000212
- [Background] Castro et al., Disease Markers Volume 2018, Article ID 4653109, 5 pages https://doi.org/10.1155/2018/4653109